CLINICAL TRIAL: NCT00065988
Title: Health Effects of Dental Amalgams in Children
Brief Title: The Children's Amalgam Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NIDCR-11886; U01DE011886 (NIH); NCT00000364 (obsolete NCT alias)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2005-08

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

INTERVENTIONS:
Device: Dispersed phase amalgam restoration /composite restoration

SUMMARY:
The Children's Amalgam Trial is one of only two randomized trials of its kind, and the only such trial in the United States, to address the potential impact of mercury exposure from amalgam restorations on neuropsychological and renal function in children.

DETAILED DESCRIPTION:
The safety of silver amalgam as a dental restorative material has been controversial since its introduction 150 years ago, but until recently it has been assumed that the exposure to mercury from dental amalgam is limited to the acute placement phase. However, some recent studies have raised safety concerns by demonstrating chronic release of mercury vapor from amalgam fillings during chewing and brushing. The Children's Amalgam Trial (CAT) is a two-arm randomized trial of safety, comparing amalgam with a mercury-free restorative material. A single masking procedure is used to ensure that all investigators and staff measuring outcomes are unaware of assigned trial arm. The study follows 534 New England children, aged 6-10 years at enrollment, for 5 years. The children were recruited from two northeastern U.S. communities, one in rural Maine, and one in urban Massachusetts. No trial subjects received prior amalgam restorations, and all were in need of at least two posterior occlusal fillings. Participants were randomized to receive either amalgam or composite material for all posterior restorations at baseline and at subsequent visits. The primary endpoint will be 5-year change in IQ scores. Secondary endpoints will include measures of other neuropsychological assessments and renal functioning.

ELIGIBILITY:
* 6 - 10 years of age at last birthday
* Fluent in English
* No prior or existing amalgam restorations
* Two or more posterior teeth with dental caries such that restoration would include the occlusal surfaces
* No clinical evidence of existing psychological, behavioral, neurologic, immunosuppressive, or renal disorders.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 534
Dates: Start 1997-09; Study Completion 2005-03

PRIMARY OUTCOMES:
IQ as measured by the WISC III Test

CONTACTS AND LOCATIONS:
Overall Officials: Sonja M McKinlay, Principal Investigator — New England Research Institutes, Inc
Locations (1):
- New England Research Institute, Watertown, Massachusetts, United States

REFERENCES:
- [Result] Bellinger DC, Trachtenberg F, Barregard L, Tavares M, Cernichiari E, Daniel D, McKinlay S. Neuropsychological and renal effects of dental amalgam in children: a randomized clinical trial. JAMA. 2006 Apr 19;295(15):1775-83. doi: 10.1001/jama.295.15.1775. PMID 16622139
- [Derived] Trachtenberg FL, Shrader P, Barregard L, Maserejian NN. Dental composite materials and renal function in children. Br Dent J. 2014 Jan;216(2):E4. doi: 10.1038/sj.bdj.2014.36. PMID 24457893
- [Derived] Maserejian NN, Hauser R, Tavares M, Trachtenberg FL, Shrader P, McKinlay S. Dental composites and amalgam and physical development in children. J Dent Res. 2012 Nov;91(11):1019-25. doi: 10.1177/0022034512458691. Epub 2012 Sep 12. PMID 22972857
- [Derived] Maserejian NN, Trachtenberg FL, Hauser R, McKinlay S, Shrader P, Bellinger DC. Dental composite restorations and neuropsychological development in children: treatment level analysis from a randomized clinical trial. Neurotoxicology. 2012 Oct;33(5):1291-7. doi: 10.1016/j.neuro.2012.08.001. Epub 2012 Aug 14. PMID 22906860
- [Derived] Maserejian NN, Trachtenberg FL, Hauser R, McKinlay S, Shrader P, Tavares M, Bellinger DC. Dental composite restorations and psychosocial function in children. Pediatrics. 2012 Aug;130(2):e328-38. doi: 10.1542/peds.2011-3374. Epub 2012 Jul 16. PMID 22802599
- [Derived] Trachtenberg F, Barregard L. Effect of storage time at -20 degrees C on markers used for assessment of renal damage in children: albumin, gamma-glutamyl transpeptidase, N-acetyl-beta-D-glucosaminidase and alpha1-microglobulin. Scand J Urol Nephrol. 2010 Nov;44(5):331-6. doi: 10.3109/00365599.2010.492785. Epub 2010 Jun 21. PMID 20560801
- [Derived] Trachtenberg F, Maserejian NN, Soncini JA, Hayes C, Tavares M. Does fluoride in compomers prevent future caries in children? J Dent Res. 2009 Mar;88(3):276-9. doi: 10.1177/0022034508330884. PMID 19329464
- [Derived] Maserejian NN, Trachtenberg F, Link C, Tavares M. Underutilization of dental care when it is freely available: a prospective study of the New England Children's Amalgam Trial. J Public Health Dent. 2008 Summer;68(3):139-48. doi: 10.1111/j.1752-7325.2007.00074.x. PMID 18248343
- [Derived] Soncini JA, Maserejian NN, Trachtenberg F, Tavares M, Hayes C. The longevity of amalgam versus compomer/composite restorations in posterior primary and permanent teeth: findings From the New England Children's Amalgam Trial. J Am Dent Assoc. 2007 Jun;138(6):763-72. doi: 10.14219/jada.archive.2007.0264. PMID 17545265